CLINICAL TRIAL: NCT02800512
Title: Robotic Sacrocolpopexy Versus High Uterosacral Ligament Suspension: A Randomized Trial
Brief Title: SCP vs HUSLS for Pelvic Organ Prolapse Repair
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 5160158
Record Dates: First submitted 2016-04-26; First posted 2016-06-15 (Estimated); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Pelvic Organ Prolapse; Cystocele; Rectocele; Enterocele
Keywords: pelvic organ prolapse; cystocele; rectocele; enterocele
MeSH Terms: conditions — Pelvic Organ Prolapse; Cystocele; Rectocele; Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacrocolpopexy (Active Comparator): Robotic sacrocolpopexy
  Interventions: Procedure: Robotic sacrocolpopexy
- HUSLS (Active Comparator): Vaginal high uterosacral ligament suspension
  Interventions: Procedure: high uterosacral ligament suspension

INTERVENTIONS:
Procedure: Robotic sacrocolpopexy — Sacrocolpopexy is a procedure to surgically correct vaginal vault prolapse where mesh is used to hold the vagina in the correct anatomical position. Robotic assistance is a minimally invasive method to perform this abdominal procedure.
  Other Names: R-SCP
  Arms: Sacrocolpopexy
Procedure: high uterosacral ligament suspension — Utilizing uterosacral ligaments to support the vaginal cuff can be performed vaginally-by passing sutures bilaterally through the uterosacral ligaments. near the level of the ischial spine. HUSLS is a vaginal minimally invasive procedure for POP.
  Other Names: HUSLS
  Arms: HUSLS

SUMMARY:
The purpose of this study is to compare the effectiveness of R-SCP versus HUSLS for treatment of pelvic organ prolapse.

DETAILED DESCRIPTION:
To compare the effectiveness of Robotic Sacrocolpopexy versus vaginal High Uterosacral Ligament Suspension for treatment of pelvic organ prolapse. Both surgeries are standard of care and are equally and widely used throughout the country with well known safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years of age or older
* Signed Informed Consent
* Symptomatic pelvic organ prolapse,
* Willing and able to complete all study visit

Exclusion Criteria:

* Non-High Uterosacral Ligament Suspension (unable to do HUSLS at time of surgery),
* Dementia or considered unable to complete questionnaires

  1. Hx of Alzheimer Disease
  2. Hx multiple strokes or other neurologic condition
  3. Caregiver states the subject is unable to complete
  4. MDs opinion
* Inability to complete follow up visits due to transportation issues

  1. No access to transportation (ie. does not have vehicle)
  2. Live > 2 hours from LLUH
  3. Does not have financial means
* Congenital anomalies

  1. Bladder Exstrophy
  2. Connective tissue disease
  3. Neovaginal prolapse
  4. Prolapse of sex change vagina
* Chronic pelvic pain

  1. > 6 months of pelvic pain of undetermined origin
  2. not cyclic pain (eg. period pain or dysmenorrhea)
  3. Patient has comorbidities of CPP
  4. Fibromyalgia
  5. Interstitial cystitis
  6. Vulvodynia
* Contraindications to Mesh,

  1. Opposition to the use mesh (ie. due to religious beliefs)
  2. History of mesh complications in past
* Pregnant or planning to become pregnant during the study period.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pelvic Organ Prolapse Quantification (pop-q) to asses change post operatively | 3 month post operative
  Pelvic organ prolapses are graded with the Pelvic Organ Prolapse Quantification (POP-Q) System.
Pelvic Organ Prolapse Quantification (pop-q) to asses change post operatively | 6 month post operative
  Pelvic organ prolapses are graded with the Pelvic Organ Prolapse Quantification (POP-Q) System.
Pelvic Organ Prolapse Quantification (pop-q) to asses change post operatively | 12 month post operative
  Pelvic organ prolapses are graded with the Pelvic Organ Prolapse Quantification (POP-Q) System.

SECONDARY OUTCOMES:
questionnaires PFDI-7 | 6 month post operative
  Subject will fill out the PFDI-7 questionnaire
questionnaires PFDI-7 | 12 month post operative
  Subject will fill out the PFDI-7 questionnaire
questionnaires PFIQ-20 | 6 month post operative
  Subject will fill out the PFIQ-20 questionnaire
questionnaires PFIQ-20 | 12 month post operative
  Subject will fill out the PFIQ-20 questionnaire
questionnaires PISQ-12 | 6 month post operative
  Subject will fill out the PISQ-12 questionnaire
questionnaires PISQ-12 | 12 month post operative
  Subject will fill out the PISQ-12 questionnaire
questionnaires PGI-I | 6 month post operative
  Subject will fill out the PGI-I
questionnaires PGI-I | 12 month post operative
  Subject will fill out the PGI-I

CONTACTS AND LOCATIONS:
Overall Officials: Sam Siddighi, Principal Investigator — Loma Linda University Health Care
Locations (1):
- Loma Linda University URO/GYN, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elliott DS, Krambeck AE, Chow GK. Long-term results of robotic assisted laparoscopic sacrocolpopexy for the treatment of high grade vaginal vault prolapse. J Urol. 2006 Aug;176(2):655-9. doi: 10.1016/j.juro.2006.03.040. PMID 16813916
- [Background] Margulies RU, Rogers MA, Morgan DM. Outcomes of transvaginal uterosacral ligament suspension: systematic review and metaanalysis. Am J Obstet Gynecol. 2010 Feb;202(2):124-34. doi: 10.1016/j.ajog.2009.07.052. PMID 20113690